CLINICAL TRIAL: NCT01359657
Title: A Phase 1b, Open-label, Multicenter Study of (BMS-936564) in Combination With Lenalidomide (Revlimid) Plus Low-dose Dexamethasone, or With Bortezomib (Velcade) Plus Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Anti-CXCR4 (BMS-936564) Alone and in Combination With Lenalidomide/Dexamethasone or Bortezomib/Dexamethasone in Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA212-002
Record Dates: First submitted 2011-05-11; First posted 2011-05-25 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ulocuplumab; Lenalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Anti-CXCR4 (BMS-936564)+Lenalidomide+Dexamethasone (Experimental)
  Interventions: Biological: Anti-CXCR4 (BMS-936564); Biological: Lenalidomide; Biological: Dexamethasone
- Arm B: Anti-CXCR4 (BMS-936564)+Bortezomib+Dexamethasone (Experimental)
  Interventions: Biological: Anti-CXCR4 (BMS-936564); Biological: Bortezomib; Biological: Dexamethasone

INTERVENTIONS:
Biological: Anti-CXCR4 (BMS-936564) — Solution, Intravenously, 1-10 mg/kg, Single 60 minute infusion once a week, 42 days (cycle 1) 28 days subsequent cycles
  Other Names: Anti-CXCR4
  Arms: Arm A: Anti-CXCR4 (BMS-936564)+Lenalidomide+Dexamethasone
Biological: Lenalidomide — Tablets, per os (by mouth route of administration) (P.O), 25 mg, daily for 21 days (Day 15-35 in cycle 1; Day 1-21 in subsequent cycles), no dosing in Cycle 1, Cycle 2 +:daily dosing from Day 1-21
  Other Names: Revlimid®
  Arms: Arm A: Anti-CXCR4 (BMS-936564)+Lenalidomide+Dexamethasone
Biological: Dexamethasone — Tablets, per os (by mouth route of administration) (P.O), 40 mg, administered with Lenalidomide once every 7 days, 42 days (cycle 1) 28 days subsequent cycles
  Arms: Arm A: Anti-CXCR4 (BMS-936564)+Lenalidomide+Dexamethasone
Biological: Anti-CXCR4 (BMS-936564) — Solution, Intravenously, 1-10 mg/kg, Single 60 minute infusion once a week, 35 days (cycle 1) 21 days subsequent cycles
  Other Names: Anti-CXCR4
  Arms: Arm B: Anti-CXCR4 (BMS-936564)+Bortezomib+Dexamethasone
Biological: Bortezomib — Intravenous (IV), 1.3 mg/m2, administered on day 15, 18, 22, 25 in cycle 1, then on Day 1, 4, 8, 11 in subsequent cycles, no dosing in Cycle 1, Cycle 2 +:dosing on Day 1, 4, 8, 11
  Other Names: Velcade®
  Arms: Arm B: Anti-CXCR4 (BMS-936564)+Bortezomib+Dexamethasone
Biological: Dexamethasone — Tablets, per os (by mouth route of administration) (P.O), 40 mg, administered on the day of (and the day after) Bortezomib infusion, 35 days (cycle 1) 21 days subsequent cycles
  Arms: Arm B: Anti-CXCR4 (BMS-936564)+Bortezomib+Dexamethasone

SUMMARY:
The purpose of this study is to determine 1) the safety and tolerability of multiple intravenous doses of anti-CXCR4 (BMS-936564) as monotherapy and as combination, and 2) the maximum tolerated dose (MTD) of BMS-936564 in combination with Lenalidomide/Dexamethasone or Bortezomib/Dexamethasone in subjects with relapsed or refractory multiple myeloma.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Subjects must have confirmed diagnosis of multiple myeloma with measurable disease Excluded are subjects with only plasmacytomas, plasma cell leukemia, or non-secretory myeloma.
* Disease must be assessed within 28 days prior to treatment initiation.
* Subjects must have evidence of relapsed or relapsed/refractory disease.
* Subjects must have received at least 2 prior regimens for multiple myeloma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2.
* Subjects must have received last treatment (ie, chemotherapy, radiotherapy, biological, immunotherapy or investigational agent [therapeutic or diagnostic]) at least 14 days prior to treatment initiation. The last treatment of systemically absorbed steroids must be at least 2 weeks or 5 half lives (whichever is shorter) before the first dose of BMS-936564.

Exclusion Criteria:

* A serious uncontrolled medical disorder or active infection.
* Current or recent (within 3 months) gastrointestinal disease or condition that could impact the absorption of orally-administered drug.
* Inability to swallow oral medication.
* Uncontrolled or significant heart disease.
* Any other malignancy, excluding basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, localized prostate cancer, or superficial bladder cancer stage 0, from which the subject has not been disease-free for at least 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose | 42 days in Arm A
Determination of maximum tolerated dose | 35 days in Arm B

SECONDARY OUTCOMES:
Safety and tolerability will be analyzed for all patients. Safety endpoints will be based on adverse event reports, and include frequent adverse event (AE)s, serious adverse event (SAE)s and lab abnormalities | Safety will be evaluated up to 2 years
  Additionally safety will be measures using vital signs, electrocardiogram (ECG)s, Multiple gated acquisition scan (MUGA) or echocardiograms (ECHO), physical examination, radiology exams, skeletal survey and clinical laboratory tests
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be maximum observed concentration (Cmax) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be trough observed concentration (Cmin) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be time of maximum observed concentration (Tmax) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be area under the concentration-time curve in one dosing interval (AUC (TAU)) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be half-life (T-Half) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be total body clearance (CLT) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Pharmacokinetic (PK) measures will be collected for all patients who received study medication. The pharmacokinetic parameters will be volume of distribution at steady-state (Vss) | PK samples will be collected multiple time points during Cycle 1 (Arm A is Day 1-42, Arm B is Day 1-35). In Cycle 2 samples will be collected on days 1, 8 & 15, at end of treatment & during the follow-up visit. Similar PK sampling will occur in Arm A & B
Individual tumor responses as defined by the International Myeloma Working Group Uniform Response Criteria (IMWG) for Multiple Myeloma (MM) will be used to monitor efficacy. For this assessment blood urine, and/or bone marrow assessment will be used | within 28 days prior to first dose
Anti-tumor response will be assessed by IMWG criteria (blood and urine; Bone marrow will not be collected unless to confirm complete response (CR)) | On Cycle 1 day 14
Anti-tumor response will be assessed by IMWG criteria (blood and urine; Bone marrow assessment will be collected during screening period, at end of cycle 1, end of cycle 4 and to confirm CR ) | At end of each Cycle
Samples will be collected to characterize immunogenicity | For Arm A, blood samples will be collected prior to dosing administration on Cycle 1 (predose & Days 1, 15, & 29), Cycle 2 Day 1, Cycle 3 Day 1; & Day 1 of Cycle 6 & every 6 cycles, end of treatment, & at 3 & 6 month follow-up visits, if available
Samples will be collected to characterize immunogenicity | For Arm B, blood samples will be collected at Cycle 1 (predose & Days 1, 15, & 29), Cycle 2 Day 1, Cycle 3 Day 1; Cycle 4 Day 1; & Day 1 on Cycle 8 & every 8 cycles, if available, end of treatment, & at 3 & 6 month follow-up visits, if available
Baseline level of cytokines/chemokines/growth factors will be determined, but not limited to SDF1 in peripheral blood and bone marrow | Sample will be collected within 28 days prior to first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University Of Kansas Cancer Center And Medical Pavillion, Westwood, Kansas
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - University Of Washington School Of Medicine, Seattle, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx